CLINICAL TRIAL: NCT02477800
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Aducanumab (BIIB037) in Subjects With Early Alzheimer's Disease
Brief Title: 221AD301 Phase 3 Study of Aducanumab (BIIB037) in Early Alzheimer's Disease
Acronym: ENGAGE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was discontinued based on futility analysis done and not based on safety concerns. Follow-up visits and closing out study activities are completed
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 221AD301; 2015-000966-72 (EudraCT Number)
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer's Disease
Keywords: BIIB037; Aducanumab
MeSH Terms: conditions — Alzheimer Disease | interventions — aducanumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose (Experimental): Monthly intravenous (IV) infusion
  Interventions: Drug: Aducanumab (BIIB037); Drug: Placebo
- High Dose (Experimental): Monthly intravenous (IV) infusion
  Interventions: Drug: Aducanumab (BIIB037); Drug: Placebo

INTERVENTIONS:
Drug: Aducanumab (BIIB037) — Low dose
  Arms: Low Dose
Drug: Aducanumab (BIIB037) — High dose
  Arms: High Dose
Drug: Placebo — Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of monthly doses of aducanumab in slowing cognitive and functional impairment as measured by changes in the Clinical Dementia Rating-Sum of Boxes (CDR-SB) score as compared with placebo in participants with early AD. Secondary objectives are to assess the effect of monthly doses of aducanumab as compared with placebo on clinical progression as measured by Mini-Mental State Examination (MMSE), AD Assessment Scale-Cognitive Subscale (13 items) [ADAS-Cog 13], and AD Cooperative Study-Activities of Daily Living Inventory (Mild Cognitive Impairment version) [ADCS-ADL-MCI].

ELIGIBILITY:
Key Inclusion Criteria:

* Must meet all of the following clinical criteria for MCI due to AD or mild AD and must have:
* A Clinical Dementia Rating (CDR)-Global Score of 0.5.
* Objective evidence of cognitive impairment at screening
* An MMSE score between 24 and 30 (inclusive)
* Must have a positive amyloid Positron Emission Tomography (PET) scan
* Must consent to apolipoprotein E (ApoE) genotyping
* If using drugs to treat symptoms related to AD, doses must be stable for at least 8 weeks prior to screening visit 1
* Must have a reliable informant or caregiver

Key Exclusion Criteria:

* Any medical or neurological condition (other than Alzheimer's Disease) that might be a contributing cause of the subject's cognitive impairment
* Have had a stroke or Transient Ischemic Attack (TIA) or unexplained loss of consciousness in the past 1 year
* Clinically significant unstable psychiatric illness in past 6 months
* History of unstable angina, myocardial infarction, advanced chronic heart failure, or clinically significant conduction abnormalities within 1 year prior to Screening
* Indication of impaired renal or liver function
* Have human immunodeficiency virus (HIV) infection
* Have a significant systematic illness or infection in past 30 days
* Relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities
* Any contraindications to brain magnetic resonance imaging (MRI) or PET scans
* Alcohol or substance abuse in past 1 year
* Taking blood thinners (except for aspirin at a prophylactic dose or less)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1653 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (178):
- United States (59):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - University of California - Los Angeles, Los Angeles, California
  - UCSF - Memory and Aging Center, San Francisco, California
  - California Neuroscience Research Medical Group Inc., Sherman Oaks, California
  - Southern California Research LLC, Simi Valley, California
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Compass Research Main, Orlando, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - USF Health Byrd Institute, Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Compass Research Main, The Villages, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Via Christi Research, a division of Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Brigham & Women's Hosp End/Dbt, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Donald S. Marks, M.D., P.C., Plymouth, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Las Vegas Medical research, Las Vegas, Nevada
  - Advanced Memory Research Institute of NJ, PC, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - New York University Medical Center PRIME, New York, New York
  - University of Rochester, Rochester, New York
  - ANI Neurology, PLLC d/b/a Alzheimer's Memory Center, Charlotte, North Carolina
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Northeastern Pennsylvania Memory and Alzheimer's Center, Plains, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Neurology Clinic, PC, Cordova, Tennessee
  - University of Tennessee Medical Center. Knoxville, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Australia (12):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Central Coast Neurosciences Research, Gosford, East Gosford, New South Wales
  - Central Coast Neurosciences Research, Erina, New South Wales
  - KARA Institute for Neurological Diseases, North Ryde, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Toowoomba Base Hospital, Toowoomba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Neurodegenerative Disorders Research, West Perth, Western Australia
- Austria (2):
  - LKH - Universitaetsklinikum Graz, Graz
  - Christian-Doppler-Klinik - Universitätsklinikum Salzburg, Salzburg
- Canada (8):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - The Medical Arts Health Research Group, Penticton, British Columbia
  - UBC Hospital, Vancouver, British Columbia
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - The Montreal Neurological Institute, Montreal, Quebec
  - McGill Centre for Studies in Aging, Verdun, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec
- Denmark (4):
  - CCBR - Ålborg - DK, Aalborg
  - CCBR - Ballerup - DK, Ballerup Municipality
  - Rigshospitalet, København Ø
  - CCBR - Vejle - DK, Vejle
- France (7):
  - Hopital Louis Pasteur Colmar, Strasbourg, Bas Rhin
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - CHU Reims - Hôpital Maison Blanche, Reims, Marne
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - Groupe hospitalier Broca - La Rochefoucauld - La Collégiale, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Germany (11):
  - Praxis Dr. Scholz, Böblingen, Baden-Wurttemberg
  - Aerztliche Gemeinschaftspraxis, Ostfildern, Baden-Wurttemberg
  - Neuro MVZ Stuttgart, Stuttgart, Baden-Wurttemberg
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt, Bavaria
  - Praxis Dr. med. Bergmann, Neuburg am Inn, Bavaria
  - Neurologische Gemeinschaftspraxis Kassel, Kassel, Hesse
  - Klinische Forschung Hannover-Mitte GmbH, Hanover, Lower Saxony
  - Universitaetsklinikum Aachen AOeR, Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Bonn AoeR, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
- Italy (13):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona, Ancona
  - Fondazione Istituto G.Giglio di Cefalù, Cefalù, Palermo
  - Azienda Ospedaliera Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Ospedale San Raffaele, Milan
  - Casa di Cura del Policlinico, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Seconda Università degli Studi di Napoli, Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (23):
  - Research Site, Chiba, Chiba
  - Research Site, Inzai-shi, Chiba
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Aizuwakamatsu-shi, Fukushima
  - Research Site, Asahikawa-shi, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Atsugi-shi, Kanagawa
  - Research Site, Kamakura-shi, Kanagawa
  - Research Site, Kawasaki-Shi, Kanagawa
  - Yokohama, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Nagaoka-shi, Niigata
  - Research Site, Iruma-gun, Saitama
  - Research Site, Kasukabe-shi, Saitama
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Bunkyō City, Tokyo-To
  - Research Site, Shinjuku-ku (I), Tokyo-To
  - Research Site, Shinjuku-ku, Tokyo-To
  - Research Site, Yamagata, Yamagata
  - Research Site, Itabashi-ku
  - Research Site, Kiyose-shi
  - Research Site, Kodaira-shi
- Portugal (6):
  - Hospital Professor Doutor Fernando Fonseca, E.P.E., Amadora
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitário de Coimbra E.P.E, Coimbra
  - CUF Alvalade, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - Campus Neurologico Senior, Torres Vedras
- South Korea (6):
  - Inha University Hospital, Incheon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
- Spain (8):
  - Policlinica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Fundacio ACE, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Clinica Ruber, Madrid
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- United Kingdom (13):
  - Southmead Hospital, Bristol, Avon
  - Re:Cognition Health Ltd, London, Greater London
  - Charing Cross Hospital, London, Greater London
  - The National Hospital for Neurology and Neurosurgery Centre, London, Greater London
  - Salford Royal, Salford, Greater Manchester
  - The University of Edinburgh, Edinburgh, Lothian Region
  - Manchester Royal Infirmary, Blackburn, Merseyside
  - The RICE Centre, Bath, Somerset
  - Glasgow Memory Clinic Ltd, Glasgow, Strathclyde
  - Stobhill ACH Hospital, Glasgow, Strathclyde
  - Ninewells Hospital, Dundee, Tayside Region
  - Newcastle University, Newcastle upon Tyne, Tyne & Wear
  - Kingshill Research Centre, Chippenham, Wiltshire

REFERENCES:
- [Derived] Loomis SJ, Miller R, Castrillo-Viguera C, Umans K, Cheng W, O'Gorman J, Hughes R, Budd Haeberlein S, Whelan CD. Genome-Wide Association Studies of ARIA From the Aducanumab Phase 3 ENGAGE and EMERGE Studies. Neurology. 2024 Feb 13;102(3):e207919. doi: 10.1212/WNL.0000000000207919. Epub 2023 Dec 28. PMID 38165296
- [Derived] Muralidharan KK, Kowalski KG, Tong X, Haeberlein SB, Rajagovindan R, Nestorov I. Characterization of exposure-Clinical Dementia Rating-Sum of Boxes relationship in subjects with early Alzheimer's disease from the aducanumab Phase 3 trials. J Pharmacokinet Pharmacodyn. 2023 Feb;50(1):45-62. doi: 10.1007/s10928-022-09839-3. Epub 2023 Jan 4. PMID 36600109
- [Derived] Salloway S, Chalkias S, Barkhof F, Burkett P, Barakos J, Purcell D, Suhy J, Forrestal F, Tian Y, Umans K, Wang G, Singhal P, Budd Haeberlein S, Smirnakis K. Amyloid-Related Imaging Abnormalities in 2 Phase 3 Studies Evaluating Aducanumab in Patients With Early Alzheimer Disease. JAMA Neurol. 2022 Jan 1;79(1):13-21. doi: 10.1001/jamaneurol.2021.4161. PMID 34807243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 169 investigational sites in Australia, Austria, Canada, Denmark, France, Germany, Italy, Japan, Portugal, Republic of Korea, Spain, Taiwan, the United Kingdom (UK) and the United States (US) from 13 August, 2015 to 04 July, 2018.
Pre-assignment Details: A total of 1653 participants with Alzheimer's disease were enrolled and randomized in the study. Of these, 1647 participants received the study drug in placebo-controlled (PC) period. After completing PC period, 852 participants entered and dosed in long-term extension (LTE) period and no participants completed the study due to early termination of the study.
Groups:
- Placebo (PC Period): Participants received a maximum of 20 infusions of BIIB037-matching placebo intravenously (IV) in PC period, administered approximately once every 4 weeks for up to approximately 1.5 years.
- BIIB037 Low Dose (PC Period): Participants received a maximum of 20 infusions of BIIB037 low dose IV in PC period, administered approximately once every 4 weeks for up to approximately 1.5 years.
- BIIB037 High Dose (PC Period): Participants received a maximum of 20 infusions of BIIB037 high dose IV in PC period, administered approximately once every 4 weeks for up to approximately 1.5 years.
- BIIB037 Late Start: Low Dose (LTE Period): Following PC period, participants randomized to placebo received BIIB037 low dose, IV infusion, approximately every 4 weeks for up to 2 years in LTE period.
- BIIB037 Late Start: High Dose (LTE Period): Following PC period, participants randomized to placebo received BIIB037 high dose, IV infusion, approximately every 4 weeks for up to 2 years in LTE period.
- BIIB037 Early Start: Low Dose (LTE Period): Following PC period, participants randomized to low dose BIIB037 continued to receive the same dose, IV infusion, approximately every 4 weeks for up to 2 years in LTE period.
- BIIB037 Early Start: High Dose (LTE Period): Following PC period, participants randomized to high dose BIIB037 continued to receive the same dose, IV infusion, approximately every 4 weeks for up to 2 years in LTE period.
Period: Placebo-Controlled Period
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period) | BIIB037 Late Start: Low Dose (LTE Period) | BIIB037 Late Start: High Dose (LTE Period) | BIIB037 Early Start: Low Dose (LTE Period) | BIIB037 Early Start: High Dose (LTE Period)
Started | 545 | 547 | 555 | 0 | 0 | 0 | 0
Completed | 325 | 325 | 288 | 0 | 0 | 0 | 0
Not Completed | 220 | 222 | 267 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 16 | 25 | 28 | 0 | 0 | 0 | 0
Not completed — Change of Treatment | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Consent Withdrawn | 26 | 16 | 27 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 3 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Relocation | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Investigator | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study Visit Burden | 5 | 3 | 11 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 5 | 3 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 161 | 161 | 189 | 0 | 0 | 0 | 0
Period: Long Term Extension Period
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period) | BIIB037 Late Start: Low Dose (LTE Period) | BIIB037 Late Start: High Dose (LTE Period) | BIIB037 Early Start: Low Dose (LTE Period) | BIIB037 Early Start: High Dose (LTE Period)
Started | 0 | 0 | 0 | 150 (12 PC completers did not enter LTE.) | 152 (11 PC completers did not enter LTE.) | 299 (26 PC completers did not enter LTE.) | 251 (37 PC completers did not enter LTE.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 150 | 152 | 299 | 251
Not completed — Adverse Event | 0 | 0 | 0 | 6 | 2 | 4 | 3
Not completed — Death | 0 | 0 | 0 | 1 | 1 | 1 | 2
Not completed — Consent Withdrawn | 0 | 0 | 0 | 10 | 4 | 13 | 16
Not completed — Disease Progression | 0 | 0 | 0 | 3 | 1 | 1 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Site Terminated By Sponsor | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Study Visit Burden | 0 | 0 | 0 | 3 | 0 | 2 | 2
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 1 | 3 | 3 | 1
Not completed — Reason not Specified | 0 | 0 | 0 | 126 | 140 | 270 | 224

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) population was defined as all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period) | Total
Number analyzed (Participants) | 545 | 547 | 555 | 1647
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (7.72) | 70.4 (6.96) | 70.0 (7.65) | 70.1 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 284 | 292 | 863
  Male | 258 | 263 | 263 | 784
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 55 | 55 | 65 | 175
  Black or African American | 5 | 1 | 2 | 8
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 1
  White | 413 | 412 | 413 | 1238
  Not Reported due to Confidentiality Regulations | 69 | 74 | 72 | 215
  Other | 3 | 4 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 13 | 37
  Not Hispanic or Latino | 489 | 492 | 499 | 1480
  Not Reported due to Confidentiality Regulations | 43 | 44 | 43 | 130

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SB) Score at Week 78
Description: CDR-SB integrates assessments from 3 domains of cognition (memory, orientation, judgment/problem-solving) and 3 domains of function (community affairs, home/hobbies, personal care). Following caregiver interview and systematic patient examination, the rater assigns a score describing the participant's current performance level in each of these domains of life functioning. Prespecified severity anchors range from none = 0, questionable = 0.5, mild = 1, moderate = 2 to severe = 3 (the personal care domain omits the 0.5 score). "Sum of boxes" scoring methodology sums the score for each of the 6 domains and provides a value ranging from 0 to 18 that can change in increments of 0.5 or greater. Higher scores indicate greater disease severity. Mixed model for repeated measures (MMRM) analysis was used to analyze change from baseline in CDR-SB. A positive change from baseline indicates clinical decline.
Time Frame: Baseline, Week 78
Population: ITT was defined as all randomized participants who had received at least one dose of study treatment (Aducanumab or Placebo). 'Number of Participants Analyzed' signifies number of participants analyzed in this outcome measure.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period)
Number analyzed (Participants) | 333 | 331 | 295
score on a scale | 1.56 (0.108) | 1.38 (0.108) | 1.59 (0.111)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB037 Low Dose (PC Period); Adjusted mean for each treatment group (Placebo, BIIB037 Low Dose, BIIB037 High Dose), difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in CDR-SB as dependent variable and with fixed effects of treatment group, categorical visit, treatment-by-visit interaction, baseline CDR-SB, baseline CDR-SB by visit interaction, baseline MMSE, AD symptomatic medication use at baseline, region, and laboratory ApoE status; Test type: Superiority; p = 0.2250, MMRM Model; Difference from Placebo = 0.110, 95% CI 2-sided [-0.469 to 0.403]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB037 High Dose (PC Period); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8330, MMRM Model; Difference from late start group = 0.03, 95% CI 2-sided [-0.262 to 0.326]

2. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Score at Week 78
Description: The MMSE is a widely used performance-based test of global cognitive status. It consists of 11 tasks that assess orientation, word recall, attention and calculation, language abilities, and visuospatial functions. The scores from the 11 tests are combined to obtain the total score, which ranges from 0 to 30, with lower scores over time indicating increasing cognitive impairment. MMRM analysis was used to analyze change from baseline in MMSE. A negative change from baseline indicates clinical decline.
Time Frame: Baseline, Week 78
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period)
Number analyzed (Participants) | 332 | 334 | 297
score on a scale | -3.5 (0.21) | -3.3 (0.21) | -3.6 (0.21)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB037 Low Dose (PC Period); Adjusted mean for each treatment group (Placebo, BIIB037 Low Dose, BIIB037 High Dose), difference from Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MMSE as dependent variable and with fixed effects of treatment group, categorical visit, treatment-by-visit interaction, baseline MMSE, baseline MMSE by visit interaction, AD symptomatic medication use at baseline, region, and laboratory ApoE status; Test type: Superiority; p = 0.4795, MMRM Model; Difference from Placebo = 0.2, 95% CI 2-sided [-0.35 to 0.74]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB037 High Dose (PC Period); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8106, MMRM Model; Difference from Placebo = -0.1, 95% CI 2-sided [-0.62 to 0.49]

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (13 Items) (ADAS-Cog 13) Score at Week 78
Description: ADAS-Cog13 comprises both cognitive tasks and clinical ratings of cognitive performance. The scale items capture word recall, ability to follow commands, the ability to correctly copy or draw an image, naming, the ability to interact with everyday objects, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure for delayed word recall and concentration/distractibility. The total score ranges from 0 to 85. An increase in score over time indicates increasing cognitive impairment. MMRM analysis was used to analyze change from baseline in ADAS-Cog 13. A positive change from baseline indicates clinical decline.
Time Frame: Baseline, Week 78
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period)
Number analyzed (Participants) | 331 | 332 | 294
score on a scale | 5.140 (0.3783) | 4.558 (0.3780) | 4.552 (0.3872)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB037 Low Dose (PC Period); Adjusted mean for each treatment group (Placebo,BIIB037 Low Dose,BIIB037 High Dose),difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in ADAS-Cog 13 as dependent variable and with fixed effects of treatment group,categorical visit,treatment-by-visit interaction,baseline ADAS-Cog 13,baseline ADAS-Cog 13 by visit interaction,baseline MMSE,AD symptomatic medication use at baseline,region,and laboratory ApoE status; Test type: Superiority; p = 0.2536, MMRM Model; Difference from Placebo = -0.583, 95% CI 2-sided [-1.5835 to 0.4181]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB037 High Dose (PC Period); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2578, MMRM Model; Difference from Placebo = -0.588, 95% CI 2-sided [-1.6067 to 0.4309]

4. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (Mild Cognitive Impairment Version) (ADCS-ADL-MCI) Score at Week 78
Description: The ADCS-ADL-MCI consists of 17 instrumental items (e.g., shopping, preparing meals, using household appliances) and 1 basic item (getting dressed). Ratings reflect caregiver observations about the patient's actual functioning over the previous month and provide an assessment of change in the functional state of the participant over time. The total score ranges from 0 to 53, with lower values over time reflecting functional deterioration. MMRM analysis was used to analyze change from baseline in ADAS-ADL-MCI. A negative change from baseline indicates clinical decline.
Time Frame: Baseline, Week 78
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period)
Number analyzed (Participants) | 331 | 330 | 298
score on a scale | -3.8 (0.35) | -3.1 (0.35) | -3.1 (0.35)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB037 Low Dose (PC Period); Adjusted mean for each group (Placebo, BIIB037 Low Dose, BIIB037 High Dose), difference with Placebo,95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in ADCS-ADL-MCI as dependent variable and with fixed effects of treatment group,categorical visit,treatment-by-visit interaction, baseline ADCS-ADL-MCI, baseline ADCS-ADL-MCI by visit interaction, baseline MMSE AD symptomatic medication use at baseline,region, and laboratory ApoE status; Test type: Superiority; p = 0.1225, MMRM Model; Difference from Placebo = 0.7, 95% CI 2-sided [-0.19 to 1.64]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB037 High Dose (PC Period); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1506, MMRM Model; Difference from late start group = 0.7, 95% CI 2-sided [-0.25 to 1.61]

ADVERSE EVENTS:
Time Frame: From First Dose to End of Study (up to 4 years)
Description: Safety population was all randomized participants who received at least one dose of study treatment. In PC period, 5 participants randomized to placebo, inadvertently received 1 or more doses of active treatment during the PC period. For participants affected, a participant was counted only once within each system organ class/preferred term/study period.
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period) | BIIB037 Late Start: Low Dose (LTE Period) | BIIB037 Late Start: High Dose (LTE Period) | BIIB037 Early Start: Low Dose (LTE Period) | BIIB037 Early Start: High Dose (LTE Period)
All-Cause Mortality (participants affected / at risk) | 0/540 | 3/549 | 2/558 | 1/150 | 1/152 | 1/299 | 2/251
Serious Adverse Events (participants affected / at risk) | 70/540 | 76/549 | 79/558 | 19/150 | 14/152 | 35/299 | 25/251
Other Adverse Events (participants affected / at risk) | 327/540 | 396/549 | 410/558 | 89/150 | 90/152 | 130/299 | 121/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PC Period) (N=540) | BIIB037 Low Dose (PC Period) (N=549) | BIIB037 High Dose (PC Period) (N=558) | BIIB037 Late Start: Low Dose (LTE Period) (N=150) | BIIB037 Late Start: High Dose (LTE Period) (N=152) | BIIB037 Early Start: Low Dose (LTE Period) (N=299) | BIIB037 Early Start: High Dose (LTE Period) (N=251)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 4 | 3 | 0 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Labyrinthine fistula (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incarcerated hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 1 | 2 | 0 | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 4 | 0 | 1 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Serratia infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 12 | 4 | 4 | 0 | 7 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 2 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood ketone body increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0 | 2 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tubular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 0 | 2 | 7 | 2 | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dementia alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dementia with lewy bodies (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dystonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Focal dyscognitive seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1
Superficial siderosis of central nervous system (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 4 | 5 | 1 | 1 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0
Vertebral artery dissection (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Persistent depressive disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychogenic tremor (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostatic dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 0 | 1 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 4 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PC Period) (N=540) | BIIB037 Low Dose (PC Period) (N=549) | BIIB037 High Dose (PC Period) (N=558) | BIIB037 Late Start: Low Dose (LTE Period) (N=150) | BIIB037 Late Start: High Dose (LTE Period) (N=152) | BIIB037 Early Start: Low Dose (LTE Period) (N=299) | BIIB037 Early Start: High Dose (LTE Period) (N=251)
Diarrhoea (Gastrointestinal disorders) | 44 | 49 | 52 | 6 | 8 | 16 | 9
Nausea (Gastrointestinal disorders) | 42 | 30 | 40 | 5 | 10 | 13 | 6
Fatigue (General disorders) | 38 | 30 | 34 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 64 | 65 | 68 | 11 | 11 | 20 | 15
Upper respiratory tract infection (Infections and infestations) | 49 | 47 | 51 | 10 | 12 | 21 | 20
Urinary tract infection (Infections and infestations) | 37 | 30 | 34 | 12 | 5 | 16 | 14
Contusion (Injury, poisoning and procedural complications) | 23 | 33 | 36 | 4 | 6 | 17 | 4
Fall (Injury, poisoning and procedural complications) | 54 | 70 | 83 | 11 | 18 | 28 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 27 | 35 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 42 | 26 | 44 | 0 | 0 | 0 | 0
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 34 | 89 | 102 | 23 | 22 | 16 | 18
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 16 | 140 | 195 | 33 | 43 | 19 | 21
Dizziness (Nervous system disorders) | 54 | 49 | 54 | 6 | 4 | 14 | 13
Headache (Nervous system disorders) | 81 | 98 | 115 | 14 | 19 | 27 | 24
Superficial siderosis of central nervous system (Nervous system disorders) | 10 | 51 | 88 | 15 | 17 | 9 | 14
Anxiety (Psychiatric disorders) | 28 | 32 | 28 | 7 | 4 | 12 | 14
Depression (Psychiatric disorders) | 34 | 40 | 34 | 8 | 5 | 9 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 29 | 19 | 9 | 4 | 12 | 6
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 5 | 9 | 4 | 3

LIMITATIONS AND CAVEATS:
The study was halted prematurely based on a prespecified futility analysis and not based on safety concerns. Participants discontinued due to study termination are included in "Reason not Specified" category in participant flow tables above.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT02477800/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02477800/SAP_001.pdf